CLINICAL TRIAL: NCT04874428
Title: Pharmacokinetics and Pharmacodynamics of Single Doses of Rivaroxaban and Apixaban in Patients With Compensated Liver Cirrhosis
Brief Title: Direct Oral Anticoagulants (Rivaroxaban and Apixaban) in Patients With Liver Cirrhosis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UVCMHEP001
Record Dates: First submitted 2021-04-30; First posted 2021-05-05 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Liver Cirrhosis
Keywords: Rivaroxaban; Apixaban; Factor Xa Inhibitors; Antithrombins; Serine Proteinase Inhibitors; Protease Inhibitors; Enzyme Inhibitors; Anticoagulants; Pharmacokinetics; Pharmacodynamics; Thromboembolism; Venous Thromboembolism; Embolism and Thrombosis; Vascular Diseases; Cardiovascular Diseases; Liver Cirrhosis; Liver Diseases
MeSH Terms: conditions — Liver Cirrhosis; Thromboembolism; Venous Thromboembolism; Embolism and Thrombosis; Vascular Diseases; Cardiovascular Diseases; Liver Diseases | interventions — Rivaroxaban; Tablets; apixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rivaroxaban (Experimental): Pharmacokinetics and pharmacodynamics of rivaroxaban
  Interventions: Drug: Rivaroxaban 10 mg Oral Tablet
- Apixaban (Experimental): Pharmacokinetics and pharmacodynamics of apixaban
  Interventions: Drug: Apixaban 2.5 mg Oral Tablet

INTERVENTIONS:
Drug: Rivaroxaban 10 mg Oral Tablet — Administration of one single dose of rivaroxaban (10 mg) in tablet form.
  Other Names: Xarelto
  Arms: Rivaroxaban
Drug: Apixaban 2.5 mg Oral Tablet — Administration of one single dose of apixaban (2.5 mg) in tablet form.
  Other Names: Eliquis
  Arms: Apixaban

SUMMARY:
The aim of this study is to investigate the pharmacokinetic and pharmacodynamic parameters of rivaroxaban and apixaban in patients with compensated liver cirrhosis (Child-Pugh class A and B).

The enrolled participants receive a prophylactic single oral dose of either rivaroxaban (10 mg) or apixaban (2.5 mg) at around 8 a.m. on the day of the trial. Blood samples are taken 0.5 hours pre-dose and 1, 2, 3, 4, 6, 8, 12 hours post-dose.

A follow-up telephone call is performed 5 days after the study intervention to collect safety data.

DETAILED DESCRIPTION:
Background:

Cirrhosis is an increasing cause of morbidity and mortality in more developed countries, being the 14th most common cause of death worldwide but fourth in central Europe. Patients with liver cirrhosis frequently require anticoagulation and the main indication for anticoagulation in cirrhotic patients is portal vein thrombosis.

The most studied and used anticoagulants for patients with liver cirrhosis so far have been low molecular weight heparins (LMWH) and warfarin (vitamin K antagonist, VKA). LMWH are safe and effective in cirrhotic patients, reduce the risk of portal vein thrombosis and liver decompensation and improve liver function and Child-Pugh score as well as overall survival. On the other side, VKA treatment is challenging in patients with liver disease as warfarin has high plasma protein binding (~99%) and is predominantly eliminated by the liver through a cytochrome P450-dependent metabolism, and INR at baseline is often elevated. Thus, the dose of warfarin and the target International Normalized Ratio (INR) are not well defined in this population. Both of them, LMWH and VKA, have some important drawbacks. On one hand, the LMWH require a daily subcutaneous injection. On the other hand, the orally ingested VKA need monitoring of the INR value. The measurement of the INR value in patients with liver cirrhosis is inadequate to guide anticoagulation as the INR value is altered in association with liver cirrhosis.

Because of the enumerated reasons above, it might be desirable to use direct oral anticoagulants (DOAC) in patients with liver cirrhosis. DOAC do not need routine INR monitoring and can be taken orally at a fixed dose and hence do not need injection. Furthermore, DOAC have a quicker onset of action than Warfarin and show a lower risk of bleeding.

The DOAC rivaroxaban and apixaban are approved for the prevention of venous thromboembolic events in patients who have undergone elective hip or knee replacement surgery, for the treatment of deep vein thrombosis (DVT) and pulmonary embolism (PE) and to prevent recurrent DVT and PE. Furthermore, they are approved for the prevention of stroke and systemic embolism in case of non-valvular atrial fibrillation. It is important to note that DOAC are already used off label in cirrhotic patients with Child Pugh class A and B. DOAC are not recommended for cirrhotic patients with Child Pugh class C.

However, the scientific evidence for the use of DOAC in cirrhotic patients is scarce as most randomized trials studying DOAC have excluded patients with remarkable liver disease and cirrhosis. Therefore, only limited data exists about the efficacy and safety of DOAC in this specific population. Nevertheless, some studies about the use of DOAC in cirrhotic patients yet exist. As it stands now, studies say it is reasonable to consider DOAC as an alternative in patients with compensated liver cirrhosis. According to them, DOAC appear to be as safe and efficacious as traditional anticoagulants in patients with compensated cirrhosis, provided that liver function is within Child-Pugh stages A or B. However, randomized trials are necessary to investigate the safety and efficacy of DOAC in more detail, especially to establish future guidelines of their use in cirrhosis.

The concerns about the use of DOAC in cirrhotic patients arise due to multiple reasons. One important point is that patients with liver cirrhosis show haemostatic alterations, which affect pro- and anticoagulant state. Affected from the haemostatic alterations are primary haemostasis, coagulation and fibrinolysis. The primary haemostasis undergoes both, prothrombotic (increased von Willebrand factor) and prohaemorrhagic (thrombocytopenia and in vitro thrombocytopathy) changes and possibly results in a rebalanced primary haemostasis. The coagulation shifts to a rather procoagulant state. The reduced activity of coagulation factors is counterbalanced by an increase in factor VIII, decrease of natural anticoagulants, complex changes in circulating microparticles, cell-free DNA and neutrophil extracellular traps. Concerning fibrinolysis, it is not yet clear whether the changes shift fibrinolysis or not. In summary, the changes overall result in a rather prothrombotic state. Another reason for concerns is, that DOAC are metabolized via the liver to various degrees. The two drugs that will be investigated in this trial, rivaroxaban and apixaban, are partially metabolized via cytochrome P450. Considering this, pharmacokinetics and pharmacodynamics of these DOAC can change according to the stage of liver cirrhosis. This could possibly lead to a shift in the risk/benefit ratio of DOAC for cirrhotic patients.

Until now, there exists no randomized trial comparing the safety and efficacy of DOAC versus traditional anticoagulants. Furthermore, as can be seen above, cirrhotic patients were excluded from most randomized trials investigating DOAC. This phase 1 clinical trial offers the opportunity to investigate pharmacokinetics and pharmacodynamics of DOAC in cirrhotic patients. The results of this trial might help to design larger trials in this specific patient population with the final goal of safe and efficient use of rivaroxaban and apixaban in patients with compensated liver cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Patient with previously diagnosed liver cirrhosis (Child-Pugh score grade A and B).
* Written informed consent

Exclusion Criteria:

* Positive pregnancy test (only for women in childbearing age with intact uterus), pregnancy or nursing women
* Intake of prophylactic or therapeutic oral anticoagulant (phenprocoumon, acenocoumarol, dabigatran etc.) 2 weeks prior to inclusion in the study
* Application of parenteral anticoagulant, e.g. unfractionated heparin, low molecular weight heparins, heparin derivatives (fondaparinux etc.) 1 week prior to inclusion in the study
* Pharmacologic platelet inhibition within 2 weeks prior to inclusion in the study
* Known coagulation disorders (e.g. von Willebrand's disease, hemophilia)
* Active, clinically significant bleeding
* Congenital or acquired bleeding disorder
* High risk of bleeding (e.g. active ulcerative gastrointestinal disease)
* Uncontrolled severe hypertension
* Vascular retinopathy
* Acute infection
* Acute bacterial endocarditis
* Severe anemia (haemoglobin ≤100 g/L)
* Hereditary galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption
* Severe liver dysfunction (Child-Pugh Score grade C)
* Hepatic encephalopathy ≥ grade 3
* Severe renal impairment with a creatinine clearance (GFR) of <30 ml/min
* Known intolerance to the study medications rivaroxaban and/or apixaban
* Concomitant treatment with a strong CYP3A4 inhibitor (e.g., ketoconazole, itraconazole, lopinavir, ritonavir, indinavir).
* Concomitant treatment with a P-glycoprotein inhibitor and a weak or moderate CYP3A4 inhibitor (e.g., erythromycin, azithromycin, diltiazem, verapamil, quinidine, ranolazine, dronedarone, amiodarone, felodipine).
* Concomitant treatment with a P-glycoprotein inducer and a strong CYP3A4 inducer (e.g., carbamazepine, phenytoin, rifampicin).
* Wash-out period of less than two weeks prior to the application of study drug in case of prior treatment with a strong CYP3A4 inhibitor or a P-glycoprotein inhibitor and weak or moderate CYP3A4 inhibitor or with a P-glycoprotein inducer or strong CYP3A4 inducer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-05-19 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) of rivaroxaban | Up to 12 hours
Maximum plasma concentration (Cmax) of rivaroxaban | Up to 12 hours
Time to maximum plasma concentration (tmax) of rivaroxaban | Up to 12 hours
Terminal half-life (t1/2) of rivaroxaban | Up to 12 hours
Trough plasma concentration (Cmin) at 24 hours post application of rivaroxaban (imputed) | 0.5 hours pre-dose
  The Cmin value at 24 hours post application is defined to be the same value measured 0.5 hours pre-dose.
AUC of apixaban | Up to 12 hours
Cmax of apixaban | Up to 12 hours
tmax of apixaban | Up to 12 hours
t1/2 of apixaban | Up to 12 hours
Cmin at 24 hours post application of apixaban (imputed) | 0.5 hours pre-dose
  The Cmin value at 24 hours post application is defined to be the same value measured 0.5 hours pre-dose.

SECONDARY OUTCOMES:
Cmax of prothrombin fragment (F1+2) after administration of rivaroxaban | Up to 12 hours
tmax of F1+2 after administration of rivaroxaban | Up to 12 hours
Cmax of thrombin-antithrombin-complexes (TAT) after administration of rivaroxaban | Up to 12 hours
tmax of TAT after administration of rivaroxaban | Up to 12 hours
Cmax of D-dimers (DD) after administration of rivaroxaban | Up to 12 hours
tmax of DD after administration of rivaroxaban | Up to 12 hours
Cmax of F1+2 after administration of apixaban | Up to 12 hours
tmax of F1+2 after administration of apixaban | Up to 12 hours
Cmax of TAT after administration of apixaban | Up to 12 hours
tmax of TAT after administration of apixaban | Up to 12 hours
Cmax of DD after administration of apixaban | Up to 12 hours
tmax of DD after administration of apixaban | Up to 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Dr. med. Guido Stirnimann, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (1):
- Department of Visceral Surgery and Medicine, University Hospital Inselspital, Berne, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tsochatzis EA, Bosch J, Burroughs AK. Liver cirrhosis. Lancet. 2014 May 17;383(9930):1749-61. doi: 10.1016/S0140-6736(14)60121-5. Epub 2014 Jan 28. PMID 24480518
- [Background] Zermatten MG, Fraga M, Moradpour D, Bertaggia Calderara D, Aliotta A, Stirnimann G, De Gottardi A, Alberio L. Hemostatic Alterations in Patients With Cirrhosis: From Primary Hemostasis to Fibrinolysis. Hepatology. 2020 Jun;71(6):2135-2148. doi: 10.1002/hep.31201. PMID 32090357
- [Background] Weinberg EM, Palecki J, Reddy KR. Direct-Acting Oral Anticoagulants (DOACs) in Cirrhosis and Cirrhosis-Associated Portal Vein Thrombosis. Semin Liver Dis. 2019 May;39(2):195-208. doi: 10.1055/s-0039-1679934. Epub 2019 Apr 12. PMID 30978730
- [Background] Elhosseiny S, Al Moussawi H, Chalhoub JM, Lafferty J, Deeb L. Direct Oral Anticoagulants in Cirrhotic Patients: Current Evidence and Clinical Observations. Can J Gastroenterol Hepatol. 2019 Jan 8;2019:4383269. doi: 10.1155/2019/4383269. eCollection 2019. PMID 30792971
- [Background] Villa E, Camma C, Marietta M, Luongo M, Critelli R, Colopi S, Tata C, Zecchini R, Gitto S, Petta S, Lei B, Bernabucci V, Vukotic R, De Maria N, Schepis F, Karampatou A, Caporali C, Simoni L, Del Buono M, Zambotto B, Turola E, Fornaciari G, Schianchi S, Ferrari A, Valla D. Enoxaparin prevents portal vein thrombosis and liver decompensation in patients with advanced cirrhosis. Gastroenterology. 2012 Nov;143(5):1253-1260.e4. doi: 10.1053/j.gastro.2012.07.018. Epub 2012 Jul 20. PMID 22819864
- [Background] Turco L, de Raucourt E, Valla DC, Villa E. Anticoagulation in the cirrhotic patient. JHEP Rep. 2019 Jul 16;1(3):227-239. doi: 10.1016/j.jhepr.2019.02.006. eCollection 2019 Sep. PMID 32039373
- [Background] De Gottardi A, Trebicka J, Klinger C, Plessier A, Seijo S, Terziroli B, Magenta L, Semela D, Buscarini E, Langlet P, Gortzen J, Puente A, Mullhaupt B, Navascues C, Nery F, Deltenre P, Turon F, Engelmann C, Arya R, Caca K, Peck-Radosavljevic M, Leebeek FWG, Valla D, Garcia-Pagan JC; VALDIG Investigators. Antithrombotic treatment with direct-acting oral anticoagulants in patients with splanchnic vein thrombosis and cirrhosis. Liver Int. 2017 May;37(5):694-699. doi: 10.1111/liv.13285. Epub 2016 Nov 19. PMID 27778440
- See also: Compendium Xarelto — https://compendium.ch/product/1111426-xarelto-filmtabl-10-mg/mpro
- See also: Compendium Eliquis — https://compendium.ch/product/1187239-eliquis-filmtabl-2-5-mg/mpro